CLINICAL TRIAL: NCT00698503
Title: M2a- 38™ Hip System Prospective Data Collection
Brief Title: A Clinical Investigation of the M2a- 38™ Hip System
Status: Terminated | Type: Observational
Why Stopped: due to low follow up
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: 12380-6
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Avascular Necrosis
Keywords: Metal on Metal; Total Hip Arthroplasty; Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- M2a- 38™ Hip System

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of the M2a- 38™ Hip System

ELIGIBILITY:
Inclusion Criteria:

* Patients having primary cemented or cementless total hip replacement for non-inflammatory degenerative joint disease (NIDJD) or any of its composite diagnosis of osteoarthritis, avascular necrosis, traumatic arthritis, subcapital fracture, legg perthes, slipped capital epiphysis, fracture of the pelvis, diastrophic variant.
* Patients with full skeletal maturity
* Patients undergoing unilateral total hip arthroplasty or bilateral total hip arthroplasty, either staged or simultaneously
* Patients of all races and gender
* Patients who are able to follow postoperative care instructions
* Patients who are able and willing to return for follow-up evaluations
* Patients have preoperative total Harris Hip Score less than 70 with at least moderate pain.

Exclusion Criteria:

* Patients diagnosed with inflammatory degenerative arthritis (IDJD) to include the following composite diagnoses: rheumatoid arthritis, systemic lupus erythematous, pigmented villonodular synovitis, juvenile rheumatoid arthritis and other arthritic processes of inflammatory or autoimmune etiology.
* Patients less than 18 years.
* Patients with the presence of a previous prosthetic hip replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.)in the hip joint to be operated.
* Patients with previous Girdlestone procedures.
* Patients with above the knee amputation of the contralateral and/or ipsilateral leg.
* Patients with osteoporosis, or marked bone loss which would preclude proper fixation of the prosthesis.
* Patients who are pregnant.
* Patients with an active or suspected infection in or around the hip.
* Patients with Parkinson's disease.
* Patients with vascular insufficiency, muscular atrophy, or neuromuscular disease in the affected limb.
* Patients with severe instability or deformity of the ligaments and/or surrounding soft tissue which would preclude stability of the prosthesis.
* Patients with a highly communicable disease or diseases that may limit follow-up (e.g. immuno-compromised conditions, hepatitis, active tuberculosis, neoplastic disease, etc.).
* Patients unwilling or unable to comply with a rehabilitation program for a cemented or cementless total hip replacement or who indicate difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patients with previous hip surgery or conditions that may interfere with the total hip replacement's survival or outcome, e.g., Paget's disease, Charcot's disease, severe osteoporosis compromising bone stock (Dorr type C bone).
* Patients who qualify for inclusion in the study, but refuse consent to participate in the study.
* Patients with a "fused" hip.
* Patients who have had a total hip arthroplasty on the contralateral hip within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have already made the decision to undergo Total Hip Replacement and will receive the M2a- 38™ Hip System
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2002-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score | 12 weeks, 1 year, 3 years, 5 years

SECONDARY OUTCOMES:
Incidence of revisions and removals | Any time

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Beres, MD, Study Director — Director, Clinical Research, Biomet Orthopedics, LLC